CLINICAL TRIAL: NCT01494012
Title: A Phase I Study Evaluating the Efficacy and Toxicity of Stereotactic Body Radiation for Metastatic or Recurrent Platinum-Resistant Ovarian Cancer
Brief Title: Phase I Stereotactic Body Radiation for Metastatic or Recurrent Platinum-Resistant Ovarian Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: low accrual
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Elizabeth Kidd, Assistant Professor of Radiation Oncology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GYNOVA0021; NCI-2011-03652 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); SU-12072011-8791 (Other: Stanford University); 22550 (Other: Stanford IRB)
Record Dates: First submitted 2011-12-13; First posted 2011-12-16 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Recurrent Ovarian Epithelial Cancer; Recurrent Ovarian Germ Cell Tumor; Malignant Tumor of Peritoneum; Stage IV Ovarian Epithelial Cancer; Stage IV Ovarian Germ Cell Tumor
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — Radiosurgery; Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (SBRT) (Experimental): Patients undergo SBRT 5 days a week for approximately 1 week in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: stereotactic body radiation therapy; Procedure: positron emission tomography; Procedure: computed tomography; Other: questionnaire administration; Drug: fludeoxyglucose F 18

INTERVENTIONS:
Radiation: stereotactic body radiation therapy — Undergo SBRT
  Other Names: SBRT; stereotactic radiation therapy; stereotactic radiotherapy
Procedure: positron emission tomography — Undergo FDG-PET/CT
  Other Names: FDG-PET; PET; PET scan; tomography, emission computed
Procedure: computed tomography — Undergo FDG-PET/CT
  Other Names: tomography, computed
Other: questionnaire administration — Ancillary studies
Drug: fludeoxyglucose F 18 — Undergo FDG-PET/CT
  Other Names: 18FDG; FDG

SUMMARY:
This phase I trial studies the side effects and the best dose of stereotactic body radiation therapy (SBRT) in treating patients with metastatic or recurrent ovarian cancer or primary peritoneal cancer. SBRT may be able to send x-rays directly to the tumor and cause less damage to normal tissue.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate response of platinum-resistant ovarian cancer to stereotactic body radiation therapy (SBRT) using fludeoxyglucose F 18 (18F-FDG) positron emission tomography (PET)/computed tomography (CT) 3 months after therapy.

II. Determine the rate of grade 3 or greater non-hematologic acute toxicity from SBRT using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

SECONDARY OBJECTIVES:

I. Evaluate response to SBRT using cancer antigen-125 (CA-125) and symptom assessment using Functional Assessment of Cancer Therapy (FACT)-Ovarian Symptom Index (FOSI).

II. Determine the rate of late and non-grade 3 acute toxicity using CTCAE version 4.0.

III. Evaluate local control, progression-free survival, and overall survival following SBRT.

OUTLINE:

Patients undergo SBRT 5 days a week for approximately 1 week in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 6 weeks, 3, 6, 9, and 12 months, and then every 6 months for 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have persistent, metastatic, or recurrent platinum resistant or refractory ovarian or primary peritoneal cancer.
* No restriction on previous treatment regimens, but patients must be at least 2 weeks out from last chemotherapy or investigational agent.
* Patients must be >= 18.
* Patients must have a life expectancy of at least 6 months.
* Patients must have KPS >= 60.
* Patients must have acceptable organ and marrow function as defined below (within 2 weeks prior to radiotherapy):

  * leukocytes >=3,000/uL
  * absolute neutrophil count >=1,500uL
  * platelets >=100,000/uL
  * total bilirubin within 1.5X normal institutional limits
  * AST(SGOT)/ALT(SGPT) <2.5 X institutional upper limit of normal
  * creatinine within normal institutional limits OR
  * creatinine clearance >=60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Patients must be willing to undergo a pre- and post-treatment FDG-PET/CT.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients should not have received radiation overlapping with the proposed treatment field.
* Patients cannot be receiving chemotherapy or other investigation agents from two weeks prior to radiation through undergoing their post-therapy FDG-PET/CT
* Patients cannot be pregnant or nursing.
* Patients cannot have disease >= 8cm or greater than 3 regions of disease.
* Patients cannot have concurrent malignancy other than non-melanoma skin cancer, non-invasive bladder cancer, or carcinoma in situ of the cervix.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-04; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Tumor response to SBRT as assessed by FDG-PET/CT | At 3 months
  FDG-PET response based on interpretation by nuclear medicine physician with measurement of the maximal standard uptake value (SUV) and identification of new sites of disease. Percentage of decreased SUVmax between the pre- and post-treatment FDG-PET/CT, evaluating means, medians, range and standard deviations.
The rate of grade 3 or greater non-hematologic acute toxicity as graded by the CTCAE v. 4.0 | 4-6 weeks, and up to 3 months after treatment
  Toxicity will be tabulated by type and grade.

SECONDARY OUTCOMES:
Measure CA-125 level | At baseline; 6 weeks; and 3, 6, and 12 months
FACT-Ovarian Symptom Index | At baseline; 6 weeks; and 3, 6, and 12 months
Late toxicity and non-grade 3 or greater acute toxicity following SBRT | At 6 weeks; 3, 6, 12, 18 and 24 months
Local control | Up to 5 years
Progression-free survival | Up to 5 years
Overall survival | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Kidd, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States